CLINICAL TRIAL: NCT04521647
Title: Effects of Menthol in E-cigarettes on Smoking Behaviors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000028570; 2U54DA036151-06 (NIH)
Record Dates: First submitted 2020-08-01; First posted 2020-08-20 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- menthol flavor (Experimental): Participants will receive 5% nicotine in an e-cigarette
  Interventions: Drug: Nicotine
- tobacco flavor (Experimental): Participants will receive 5% nicotine in an e-cigarette
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Participants will receive two nicotine concentrations via e-cigarettes. Each exposure will be 10 3-sec puffs and ad libitum use

SUMMARY:
The overall goal of this proposal is to understand the relationship between nicotine metabolism and menthol flavor in e-cigarettes on smoking behavior in smokers.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Able to read and write English.
* Smoking at least 1 menthol cigarettes/cigars/little cigars per day
* Report regular menthol cigarette use
* Have at least 200ng/ml urine cotinine
* Willing to abstain from combustible tobacco products 12 hrs prior to each experimental session.
* not planning a smoking quit attempt.
* Have not stopped use due to COVID.
* used e-cigarettes at least 10 times in the past six months.
* Fully vaccinated against COVID-19.
* must report history of JUUL and other nicotine salt/pod devices (i.e., JUUL-like)

Exclusion Criteria:

* Use of psychoactive drugs including anxiolytics, antidepressants, and other psychostimulants unless prescribed and stable for two months.
* Current diagnosis of any severe psychiatric disorder
* Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, pulmonary or hepatic pathology that would increase risk or would interfere with/mimic tobacco abstinence.
* Known hypersensitivity to propylene glycol and nut allergies.
* Pregnant or lactating females.
* current criteria for moderate or severe cannabis and alcohol use disorder per DSM-5 criteria.
* current criteria for other substance use disorders per DSM-5 criteria.
* Seeking treatment to stop smoking.
* individuals who do not want to use e-cigarettes.
* Uncontrolled asthma (defined as <20 on Asthma Control Test) AND/OR endorsement of "yes" to environmentally induced bronchospasm that requires prescription Epipen)
* blood pressure >170/>100 and heart rate >100
* vaping of CBD/THC or marijuana related products in the past 3 months
* For current THC vapers: Any report of mild or great EVALI-related symptoms (i.e. cough, shortness of breath, chest pain, nausea, vomiting, stomach pain, diarrhea, fever, chills, or weight loss) without non-EVALI reasonable and proximal cause

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine levels | up to 3 weeks
  blood samples obtained at baseline and 2, 5, 15, 30, 45, 60, 90, 120, and 180 minutes after nicotine exposure
Nicotine Metabolic Rate | up to 3 weeks
  blood samples obtained at baseline and 2, 5, 15, 30, 45, 60, 90, 120, and 180 minutes after nicotine exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States